CLINICAL TRIAL: NCT06878768
Title: Imagerie Cardiaque Ciné Par Résonance Magnétique En Respiration Libre
Brief Title: Translational Research GRICS-CineCardiac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C10-04; 2010-A00789-30 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-02-21; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Feasibility of GRICS CardioCine on Patients with Ischemic or Dilated Cardiopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Patients (Experimental)
  Interventions: Device: Additional free breathing MR acquisitions

INTERVENTIONS:
Device: Additional free breathing MR acquisitions

SUMMARY:
This project is a pilot study which aims at showing the feasibility of free breathing cardiac MRI using GRICS (Generalized Reconstruction by Inversion of Coupled System)software in a clinical environment.

The GRICS technique has been developed by the IADI (Diagnostic, Adaptive and Interventional Imaging)lab, Nancy, France. It enables free breathing MRI thanks to a reconstruction algorithm which provides artefact-free images based on raw MR data and physiological data from external sensors (respiratory belts, ECG.

In this study, we want to acquire free breathing cardiac cine images during a standard cardiac MR exam and compare those data with the breath-hold ones.

ELIGIBILITY:
Inclusion Criteria:

* candidate to cardiac MR exam because of ischemic or dilated cardiopathy
* legally an adult
* having heath insurance
* having signed the consent form

Exclusion Criteria:

* dyspnea
* atrial fibrillation
* pain while lying on the back for a long time
* inability to follow a procedure
* contraindication to MRI
* contraindication to gadolinium chelate injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Qualitative image reading by the radiologist | 1 Month
  Feasibility of GRICS CardioCine : the radiologist responds to a questionnaire
Quantitative image analysis by the radiologist | 1 Month
  Feasibility of GRICS CardioCine : the radiologist responds to a questionnaire

SECONDARY OUTCOMES:
Right ventricular end-diastolic volume | Day 1
  Free-breathing and breath-hold measurements
Left ventricular end-diastolic volume | Day 1
  Free-breathing and breath-hold measurements
Right ventricular end-systolic volume | Day 1
  Free-breathing and breath-hold measurements
Left ventricular end-systolic volume | Day 1
  Free-breathing and breath-hold measurements
Right ventricular systolic ejection volume | Day 1
  Free-breathing and breath-hold measurements
Left ventricular systolic ejection volume | Day 1
  Free-breathing and breath-hold measurements
Right ventricular ejection fractions | Day 1
  Free-breathing and breath-hold measurements
Left ventricular ejection fractions | Day 1
  Free-breathing and breath-hold measurements
Left ventricular mass in diastole | Day 1
  Free-breathing and breath-hold measurements
Aortic flow | Day 1
  Free-breathing and breath-hold measurements
Analysis of the segmental kinetics of the left ventricle | Day 1
  Free-breathing and breath-hold measurements

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided